CLINICAL TRIAL: NCT00561964
Title: Randomized, Parallel, Comparison, Double-Blind Efficacy & Safety Study of APROVEL Versus Placebo in Chinese Patients With Hypertensive Type II Diabetic Patients With Microalbuminuria
Acronym: PRIME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L_9079
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Irbesartan
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Irbesartan — Irbesartan capsules strength 150 mg. Irbesartan group will be initiated at one irbesartan and one placebo for 2 weeks and titrated at two capsules if well tolerated after 2 weeks , this dose will be maintained throughout the study without further dose-adjustment (2 capsules daily in the morning will be taken from randomization to study end)
  Arms: 1
Drug: placebo — Placebo group: 2 placebo capsules daily as a single morning intake
  Arms: 2

SUMMARY:
To evaluate the effects and safety of irbesartan on proteinuria in hypertensive patients with type Ⅱdiabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose of untreated type II diabetes mellitus patients greater than or equal to 7.0 mmol/L, or the time between diagnosis of type II diabetes mellitus and treatment > 3 months
* The patients of normal BP, or hypertensive patients receiving antihypertensive medication, Seated systolic blood pressure (SeSBP) is between 120-180mmHg and the Seated diastolic blood pressure (SeDBP) is between 80-110mmHg;
* Evidence of albuminuria defined as an AER of 20 and 500 ug/minute on a single timed overnight collection. Before randomization the patient must quality with two AERs of 3 days intervals in the absence of confounding factors such as urinary tract infection, acute febrile illness and cardiac failure. The two AERs measurement should be in the above defined range and the variability between the two AERs measurement must be <35%. Value of basal AER is calculated as the mean of the 2 measurements. The UAER measured using immunity nephelometer method (DCA2000);
* Serum creatinine < 150umol/L(1.7mg/dl) and serum potassium in the normal lab range (3.5-5.5 mol/L);
* 18 Kg/m2less than or equal to BMI less than or equal to 35Kg/m2

Exclusion Criteria:

* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2004-01; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Urine albumin excretion rate (UAER) | during the study conduct

SECONDARY OUTCOMES:
SeSBP, SeDBP, Total cholesterol, Triglycerides, HDL cholesterol, LDL cholesterol , glycated hemoglobin | during the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Martin Thoenes, Study Director — Sanofi